CLINICAL TRIAL: NCT03568890
Title: Short-Term Anticoagulation Versus Antiplatelet Therapy for Preventing Device Thrombosis Following Left Atrial Appendage Closure. The ANDES Trial
Brief Title: Short-Term Anticoagulation Versus Antiplatelet Therapy for Preventing Device Thrombosis Following Left Atrial Appendage Closure
Acronym: ANDES
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Josep Rodes-Cabau, Principal Investigator, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANDES
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Left Atrial Appendage Closure; Thrombosis; Stroke; TIA; Bleeding
Keywords: Left Atrial Appendage Closure; Anticoagulation therapy; Antiplatelet therapy
MeSH Terms: conditions — Thrombosis; Stroke; Hemorrhage | interventions — Rivaroxaban; Dabigatran; apixaban; edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anticoagulation therapy (Active Comparator): Direct oral anticoagulants (rivaroxaban, dabigatran, apixaban, or edoxaban; with dosage according to guideline recommendations) for 60 days.
  Interventions: Drug: Rivaroxaban, dabigatran, apixaban, or edoxaban
- Antiplatelet therapy (Active Comparator): Dual antiplatelet therapy with clopidogrel -75 mg/day- and low dose aspirin -80 to 125 mg/day for 60 days.
  Interventions: Drug: Clopidogrel -75 mg/day; Drug: Low dose aspirin -80 to 125 mg/day-

INTERVENTIONS:
Drug: Rivaroxaban, dabigatran, apixaban, or edoxaban — Duration of treatment: 60 days
  Arms: Anticoagulation therapy
Drug: Clopidogrel -75 mg/day — Duration of treatment: 60 days
  Arms: Antiplatelet therapy
Drug: Low dose aspirin -80 to 125 mg/day- — Duration of treatment: 60 days
  Arms: Antiplatelet therapy

SUMMARY:
The objective of the study is to compare short-term (8 weeks) anticoagulation therapy (DOAC) vs. antiplatelet therapy for the prevention of device thrombosis following transcatheter LAAC.

DETAILED DESCRIPTION:
Transcatheter left atrial appendage closure (LAAC) has emerged as an alternative to anticoagulation for preventing thromboembolic events in patients with atrial fibrillation. Whereas most complications associated with LAAC have decreased over time, the occurrence of device thrombosis remains a concern, with an incidence of 1 to 17%. Antithrombotic therapy for preventing device thrombosis following LAAC has evolved empirically, with antiplatelet therapy being the most commonly prescribed treatment. However, the rates of device thrombosis post-LAAC remain relatively high and have not decreased over time despite of increasing operator/center experience and the arrival of newer generation devices. This is of particular concern if we consider that LAAC is a preventive treatment. Experimental and mechanistic studies have suggested enhanced thrombin generation (and not platelet activation) within the days-weeks following the procedure as the most important mechanism involved in device thrombosis and appropriate short-term anticoagulation therapy with DOAC should translate into a significant reduction in the rate of device thrombosis post-LAAC.

Therefore, the objective of the study is to compare short-term (60 days) anticoagulation therapy (DOAC) vs. antiplatelet therapy for the prevention of device thrombosis following transcatheter LAAC.

It is estimated that 350 patients will take part in the study.

Update: A blinded interim analysis was performed with the analysis of clinical and TEE (central echo core lab) data from the initial 155 patients included in the study. Based on the results of the interim analysis, and considering the total number of events and the high rate (20%) of patients with either early cessation of the allocated treatment (before the 60-day TEE examination) or missing TEE at 60 days, it was decided to increase the sample size by 160 patients up to a total of 510 patients. This would ensure to include at least 350 patients with a TEE examination performed while receiving the allocated antithrombotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Successful transcatheter LAAC with any approved device
* Age≥18 years old

Exclusion Criteria:

* Absolute contraindications for anticoagulation therapy
* Absolute contraindications for antiplatelet therapy
* End-stage renal disease (CrCl <15 ml/min)
* Recent percutaneous revascularization with drug-eluting stents requiring dual antiplatelet therapy
* Prior intracranial hemorrhage
* Contraindications for TEE
* Severe pericardial effusion within the first 24 hrs following LAAC
* Major/life-threatening bleeding event within the month prior to LAAC
* Multiple bleeding events (minor or major) within the month prior to LAAC
* Major/life-threatening bleeding within the first 24 hrs following LAAC

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Device thrombosis (efficacy outcome) | 60 days after LAAC
  Evaluated by TEE
Combined outcome of all-cause mortality, bleeding, stroke, or Device thrombosis (Safety outcome) | 60 days after LAAC
  Clinically evaluated and diagnosed by the center investigators and determining a treatment change.

SECONDARY OUTCOMES:
Device thrombosis | 12 months after LAAC
  Evaluated by TEE or computed tomography
Ischemic events | 60 days, 12-month, 2-year, 3-year, 4-year and 5-year follow-up
  Stroke, TIA
Bleeding events | 60 days and 12-month, 2-year, 3-year, 4-year and 5-year follow-up
Major or Life-threatening bleeding events | 60 days and 12-month, 2-year, 3-year, 4-year and 5-year follow-up
Mortality | 60 days and 12-month, 2-year, 3-year, 4-year and 5-year follow-up
  All cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Josep Rodes-Cabau, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Asmarats L, Rodes-Cabau J. Percutaneous Left Atrial Appendage Closure: Current Devices and Clinical Outcomes. Circ Cardiovasc Interv. 2017 Nov;10(11):e005359. doi: 10.1161/CIRCINTERVENTIONS.117.005359. PMID 29146668
- [Background] Main ML, Fan D, Reddy VY, Holmes DR, Gordon NT, Coggins TR, House JA, Liao L, Rabineau D, Latus GG, Huber KC, Sievert H, Wright RF, Doshi SK, Douglas PS. Assessment of Device-Related Thrombus and Associated Clinical Outcomes With the WATCHMAN Left Atrial Appendage Closure Device for Embolic Protection in Patients With Atrial Fibrillation (from the PROTECT-AF Trial). Am J Cardiol. 2016 Apr 1;117(7):1127-34. doi: 10.1016/j.amjcard.2016.01.039. Epub 2016 Feb 1. PMID 26993976
- [Background] Saw J, Tzikas A, Shakir S, Gafoor S, Omran H, Nielsen-Kudsk JE, Kefer J, Aminian A, Berti S, Santoro G, Nietlispach F, Moschovitis A, Cruz-Gonzalez I, Stammen F, Tichelbacker T, Freixa X, Ibrahim R, Schillinger W, Meier B, Sievert H, Gloekler S. Incidence and Clinical Impact of Device-Associated Thrombus and Peri-Device Leak Following Left Atrial Appendage Closure With the Amplatzer Cardiac Plug. JACC Cardiovasc Interv. 2017 Feb 27;10(4):391-399. doi: 10.1016/j.jcin.2016.11.029. PMID 28231907
- [Background] Tzikas A, Shakir S, Gafoor S, Omran H, Berti S, Santoro G, Kefer J, Landmesser U, Nielsen-Kudsk JE, Cruz-Gonzalez I, Sievert H, Tichelbacker T, Kanagaratnam P, Nietlispach F, Aminian A, Kasch F, Freixa X, Danna P, Rezzaghi M, Vermeersch P, Stock F, Stolcova M, Costa M, Ibrahim R, Schillinger W, Meier B, Park JW. Left atrial appendage occlusion for stroke prevention in atrial fibrillation: multicentre experience with the AMPLATZER Cardiac Plug. EuroIntervention. 2016 Feb;11(10):1170-9. doi: 10.4244/EIJY15M01_06. PMID 25604089
- [Background] Lempereur M, Aminian A, Freixa X, Gafoor S, Kefer J, Tzikas A, Legrand V, Saw J. Device-associated thrombus formation after left atrial appendage occlusion: A systematic review of events reported with the Watchman, the Amplatzer Cardiac Plug and the Amulet. Catheter Cardiovasc Interv. 2017 Nov 1;90(5):E111-E121. doi: 10.1002/ccd.26903. Epub 2017 Feb 1. PMID 28145040
- [Background] Fauchier L, Cinaud A, Brigadeau F, Lepillier A, Pierre B, Abbey S, Fatemi M, Franceschi F, Guedeney P, Jacon P, Paziaud O, Venier S, Deharo JC, Gras D, Klug D, Mansourati J, Montalescot G, Piot O, Defaye P. Device-Related Thrombosis After Percutaneous Left Atrial Appendage Occlusion for Atrial Fibrillation. J Am Coll Cardiol. 2018 Apr 10;71(14):1528-1536. doi: 10.1016/j.jacc.2018.01.076. PMID 29622159
- [Background] O'Hara C, O'Hara GE, Jacques F, Champagne J, Lemyre M, Charbonneau L, O'Connor K, Bernier M, Beaudoin J, Rodes-Cabau J, Paradis JM. Run With the Hare and Hunt With the Hounds: Watchman Device Surgical Resection in the Setting of Recurrent Device Related Thrombi in a Patient With Bleeding Diathesis. JACC Cardiovasc Interv. 2016 Dec 12;9(23):e223-e225. doi: 10.1016/j.jcin.2016.09.041. No abstract available. PMID 27931603
- [Background] Rodriguez-Gabella T, Nombela-Franco L, Regueiro A, Jimenez-Quevedo P, Champagne J, O'Hara G, Bernier M, Macaya C, Rodes-Cabau J. Single Antiplatelet Therapy Following Left Atrial Appendage Closure in Patients With Contraindication to Anticoagulation. J Am Coll Cardiol. 2016 Oct 25;68(17):1920-1921. doi: 10.1016/j.jacc.2016.08.016. No abstract available. PMID 27765196
- [Background] Jalal Z, Dinet ML, Combes N, Pillois X, Renou P, Sibon I, Iriart X, Thambo JB. Percutaneous left atrial appendage closure followed by single antiplatelet therapy: Short- and mid-term outcomes. Arch Cardiovasc Dis. 2017 Apr;110(4):242-249. doi: 10.1016/j.acvd.2016.09.006. Epub 2017 Jan 3. PMID 28065447
- [Background] Rodes-Cabau J, O'Hara G, Paradis JM, Bernier M, Rodriguez-Gabella T, Regueiro A, O'Connor K, Beaudoin J, Puri R, Cote M, Champagne J. Changes in Coagulation and Platelet Activation Markers Following Transcatheter Left Atrial Appendage Closure. Am J Cardiol. 2017 Jul 1;120(1):87-91. doi: 10.1016/j.amjcard.2017.03.253. Epub 2017 Apr 12. PMID 28495432
- [Background] Schwartz RS, Holmes DR, Van Tassel RA, Hauser R, Henry TD, Mooney M, Matthews R, Doshi S, Jones RM, Virmani R. Left atrial appendage obliteration: mechanisms of healing and intracardiac integration. JACC Cardiovasc Interv. 2010 Aug;3(8):870-7. doi: 10.1016/j.jcin.2010.04.017. PMID 20723861
- [Background] Bass JL. Transcatheter occlusion of the left atrial appendage--experimental testing of a new Amplatzer device. Catheter Cardiovasc Interv. 2010 Aug 1;76(2):181-5. doi: 10.1002/ccd.22536. PMID 20665856
- [Background] Kar S, Hou D, Jones R, Werner D, Swanson L, Tischler B, Stein K, Huibregtse B, Ladich E, Kutys R, Virmani R. Impact of Watchman and Amplatzer devices on left atrial appendage adjacent structures and healing response in a canine model. JACC Cardiovasc Interv. 2014 Jul;7(7):801-9. doi: 10.1016/j.jcin.2014.03.003. PMID 25060026
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; ACC/AHA Task Force Members. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines and the Heart Rhythm Society. Circulation. 2014 Dec 2;130(23):2071-104. doi: 10.1161/CIR.0000000000000040. Epub 2014 Mar 28. No abstract available. PMID 24682348
- [Background] Verheugt FW, Granger CB. Oral anticoagulants for stroke prevention in atrial fibrillation: current status, special situations, and unmet needs. Lancet. 2015 Jul 18;386(9990):303-10. doi: 10.1016/S0140-6736(15)60245-8. Epub 2015 Mar 14. Erratum In: Lancet. 2015 Jul 18;386(9990):248. doi: 10.1016/S0140-6736(15)61114-X. PMID 25777666
- [Background] Lopez-Lopez JA, Sterne JAC, Thom HHZ, Higgins JPT, Hingorani AD, Okoli GN, Davies PA, Bodalia PN, Bryden PA, Welton NJ, Hollingworth W, Caldwell DM, Savovic J, Dias S, Salisbury C, Eaton D, Stephens-Boal A, Sofat R. Oral anticoagulants for prevention of stroke in atrial fibrillation: systematic review, network meta-analysis, and cost effectiveness analysis. BMJ. 2017 Nov 28;359:j5058. doi: 10.1136/bmj.j5058. PMID 29183961
- [Derived] Rodes-Cabau J, Nombela-Franco L, Cruz-Gonzalez I, Hibbert B, Freixa X, Masson JB, Ibrahim R, Estevez-Loureiro R, Millan X, Kass M, Paradis JM, Champagne J, Salinas P, Laffond A, Abdel-Razek O, Labinaz M, Cepas-Guillen P, Arzamendi D, Vidal-Cales P, Pavesi M, Cote M, O'Hara G, Salaun E. Short-Term Anticoagulation Versus Dual Antiplatelet Therapy for Preventing Device Thrombosis Following Left Atrial Appendage Closure: The ANDES Randomized Clinical Trial. Circulation. 2025 Dec 23;152(25):1759-1768. doi: 10.1161/CIRCULATIONAHA.125.077469. Epub 2025 Oct 26. PMID 41139402